CLINICAL TRIAL: NCT02947828
Title: Polyneuropathy in Diabetes Mellitus Type 2
Status: Completed | Type: Observational
Sponsor: Danish Pain Research Center (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IDNC-DD2-NP
Record Dates: First submitted 2016-10-25; First posted 2016-10-28 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus Type 2 Without Complication; Polyneuropathies, Diabetic; Diabetes Complications; Diabetic Peripheral Neuropathy; Chronic Pain
Keywords: Diabetes Mellitus, Type 2; Polyneuropathies, Diabetic
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Complications; Chronic Pain; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skin punch biopsies and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- T2D patients: 600 type 2 diabetes (T2D) patients recruited from the DD2 cohort
- Gender- and age-matched healthy controls: 100 healthy subjects

SUMMARY:
This is a population-based study of type 2 diabetes patients with and without neuropathy recruited from the Danish National Type 2 Diabetes cohort (DD2).

Perspective: The study will identify risk factors for developing diabetic polyneuropathy and painful diabetic polyneuropathy and provide information on the underlying mechanisms, which will hopefully contribute to significant improvements in the treatment and prevention of diabetic polyneuropathy in future.

DETAILED DESCRIPTION:
Diabetic polyneuropathy is one of the most common long-term complications of diabetes. Neuronal hyperexcitability is thought to be a key factor in the development of neuropathic pain.

The overall purpose of this study is to evaluate the prevalence and underlying mechanisms of diabetic polyneuropathy and painful diabetic polyneuropathy.

ELIGIBILITY:
Inclusion Criteria T2D patients:

* Clinical diagnosis of type 2 diabetes

Exclusion Criteria:

* Pregnancy
* Poor or no Danish language skills
* Insufficient mental capacity to provide informed consent or complete questionnaires

Additional criteria for healthy controls:

* Any neurological or psychiatric disorder
* Chronic pain
* Severe illness
* Pain treatment 3 days before the examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes patients
Sampling Method: Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Presence of diabetic polyneuropathy | 5 hours
  For case definition of neuropathy, Tesfaye et al. 2010 will be used.
Presence of painful diabetic polyneuropathy | 5 hours
  Neuropathic pain grading system. Finnerup et al. 2016 will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Sif Gylfadottir, MD, Principal Investigator — Aarhus University and Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Danish Pain Research Center, Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Yes
Data is shared among collaborators.

REFERENCES:
- [Background] Tesfaye S, Boulton AJ, Dyck PJ, Freeman R, Horowitz M, Kempler P, Lauria G, Malik RA, Spallone V, Vinik A, Bernardi L, Valensi P; Toronto Diabetic Neuropathy Expert Group. Diabetic neuropathies: update on definitions, diagnostic criteria, estimation of severity, and treatments. Diabetes Care. 2010 Oct;33(10):2285-93. doi: 10.2337/dc10-1303. PMID 20876709
- [Background] Finnerup NB, Haroutounian S, Kamerman P, Baron R, Bennett DLH, Bouhassira D, Cruccu G, Freeman R, Hansson P, Nurmikko T, Raja SN, Rice ASC, Serra J, Smith BH, Treede RD, Jensen TS. Neuropathic pain: an updated grading system for research and clinical practice. Pain. 2016 Aug;157(8):1599-1606. doi: 10.1097/j.pain.0000000000000492. PMID 27115670